CLINICAL TRIAL: NCT01791127
Title: Safety and Performance Study of the Siello S Pacing Lead
Acronym: SIELLO
Status: Terminated | Type: Observational
Why Stopped: On April 15, 2019, BIOTRONIK received FDA approval to transition the ongoing SIELLO Post Approval Registry to a new EP PASSION real-world data methodology.
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: G110221
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Safety and Effectiveness of the Siello S Lead

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pacemaker Therapy: Patients with a market-released BIOTRONIK pacemaker system including one or two Siello S leads.
  Interventions: Device: market-released BIOTRONIK pacemaker system including one or two Siello S leads.

INTERVENTIONS:
Device: market-released BIOTRONIK pacemaker system including one or two Siello S leads.

SUMMARY:
The objective of the SIELLO study is to demonstrate the safety and effectiveness of the BIOTRONIK Siello S pacing lead.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for de novo implantation of a BIOTRONIK pacemaker system, including one or two Siello S leads. Candidate meets recommendation for pacemaker system implant put forth by guidelines of relevant professional societies.
* Able to understand the nature of the study and provide informed consent.
* Available for follow-up visits on a regular basis at the investigational site for the expected 5 years of follow-up.
* Age greater than or equal to 18 years.

Exclusion Criteria:

* Enrolled in any other investigational clinical study.
* Currently implanted with a pacemaker or ICD device.
* Planned cardiac surgical procedures or interventional measures within the next 6 months.
* Expected to receive a heart transplant within 1 year.
* Life expectancy less than 1 year.
* Presence of another life-threatening, underlying illness separate from their cardiac disorder.
* Pregnant at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected for participation should be from the investigators' general patient population according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1758 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (53):
  - La Jolla, California
  - La Mesa, California
  - New Haven, Connecticut
  - Stamford, Connecticut
  - Plantation, Florida
  - St. Petersburg, Florida
  - Cumming, Georgia
  - Chicago, Illinois
  - Jerseyville, Illinois
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - Valparaiso, Indiana
  - Iowa City, Iowa
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Grand Blanc, Michigan
  - Warren, Michigan
  - Ypsilanti, Michigan
  - Tupelo, Mississippi
  - Cape Girardeau, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Bridgewater, New Jersey
  - Haddon Heights, New Jersey
  - Flushing, New York
  - Concord, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Middletown, Ohio
  - Steubenville, Ohio
  - Toledo, Ohio
  - Philadelphia, Pennsylvania
  - Wynnewood, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Lancaster, South Carolina
  - Rock Hill, South Carolina
  - West Columbia, South Carolina
  - Alice, Texas
  - Bedford, Texas
  - Orange, Texas
  - San Antonio, Texas
  - Victoria, Texas
  - Salt Lake City, Utah
  - Fredericksburg, Virginia
  - Richmond, Virginia
  - Milwaukee, Wisconsin
  - Cheyenne, Wyoming

REFERENCES:
- [Derived] Mullane S, Hicks JB, Sharmin K, Harrell C, Rock A, Miller C. Validation and Final Results from the First Cardiac Lead Post-Approval Study Using Real-World Data. Pragmat Obs Res. 2024 Dec 19;15:233-241. doi: 10.2147/POR.S499248. eCollection 2024. PMID 39720009

RESULTS

PARTICIPANT FLOW:
Groups:
- BIOTRONIK Siello S Lead: Patients with a BIOTRONIK pacemaker system including one or two Siello S leads.
Period: Overall Study
Arm/Group | BIOTRONIK Siello S Lead
Started | 1758
Completed | 286
Not Completed | 1472
Not completed — Death | 356
Not completed — Patient has withdrawn from study | 293
Not completed — Lost to Follow-up | 42
Not completed — All Siello leads are explanted | 31
Not completed — Completion of 30 day safety registry | 1
Not completed — Study terminated for EP Passion | 749

BASELINE CHARACTERISTICS:
Arm/Group | BIOTRONIK Siello S Lead
Number analyzed (Participants) | 1758
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 821
  Male | 937
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1380
  Black or African American | 112
  Hispanic or Latino | 47
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 2
  American Indian or Alaska Native | 2
  Not Reported | 193
Region of Enrollment [Number; unit: participants]
  United States | 1758
Weight [Mean (Standard Deviation); unit: pounds] — Population: Baseline characteristics are provided when available, subjects without available baseline characteristics are not included in the number of participants analyzed in this section.
  pounds
    number analyzed (Participants) | 1752
    (all) | 187.8 (51.6)
Height [Mean (Standard Deviation); unit: inches] — Population: Baseline characteristics are provided when available, subjects without available baseline characteristics are not included in the number of participants analyzed in this section.
  inches
    number analyzed (Participants) | 1749
    (all) | 66.9 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Atrial Siello S Lead Safety at 12 Months
Description: The overall percentage subjects with adverse events that require additional invasive intervention to resolve, related to the Siello leads implanted in the atrium with a BIOTRONIK Evia pacemaker device through 12 months follow-up. This was evaluated as an adverse event free-rate (AEFR).
Time Frame: 12 month
Population: The Pre-Market cohort was defined as the population of subjects who were implanted (or had an implant attempt) of an atrial Siello lead on or before the implant date of the last subject to reach the 12-month follow-up time point as of April 3, 2015 and/or experienced a qualifying event.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- BIOTRONIK Siello S Atrial Lead: Patients in the pre-market cohort with a BIOTRONIK pacemaker system including a Siello S atrial lead.
Arm/Group | BIOTRONIK Siello S Atrial Lead
Number analyzed (Participants) | 450
percentage of participants | 100 [99.2 to 100]
Statistical Analysis 1: Comparison: BIOTRONIK Siello S Atrial Lead; Test type: Superiority — The primary endpoint 1 hypothesis was evaluated by performing an exact, binomial test comparing a binomial proportion (AEFR at 12 months) to 94.0%, with Type I error (alpha) or 0.025 and power of 80%; p < 0.0001, Exact, binomial

2. Primary Outcome: Ventricular Siello S Lead Safety at 12 Months
Description: The overall percentage of subjects with adverse events that require additional invasive intervention to resolve, related to the Siello leads implanted in the ventricle with a BIOTRONIK Evia pacemaker device through 12 months follow-up. This was evaluated as an adverse event free-rate (AEFR).
Time Frame: 12-month
Population: The Pre-Market cohort was defined as the population of subjects who were implanted (or had an implant attempt) of a ventricular Siello lead on or before the implant date of the last subject to reach the 12-month follow-up time point as of April 3, 2015 and/or experienced a qualifying event.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- BIOTRONIK Siello S Ventricular Lead: Patients in the pre-market cohort with a BIOTRONIK pacemaker system including a Siello S ventricular lead.
Arm/Group | BIOTRONIK Siello S Ventricular Lead
Number analyzed (Participants) | 525
percentage of participants | 99.62 [98.6 to 100]
Statistical Analysis 1: Comparison: BIOTRONIK Siello S Ventricular Lead; The primary endpoint 2 hypothesis was evaluated by performing an exact, binomial test comparing a binomial proportion (AEFR at 12 months) to 94.0%, with Type I error (alpha) or 0.025 and power of 80%; Test type: Superiority; p < 0.0001, Exact, binomial

3. Primary Outcome: Siello S Lead Effectiveness at 12 Months
Description: Success rate of the implanted system to sense and deliver pacing at 12-months post implant.
Time Frame: 12-months
Population: The Pre-Market cohort was defined as the population of subjects who were implanted (or had an implant attempt) of one or more Siello leads on or before the implant date of the last subject to reach the 12-month follow-up time point as of April 3, 2015 and/or experienced a qualifying event.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- BIOTRONIK Siello S Lead: Patients in the pre-market cohort with a BIOTRONIK pacemaker system including one or two Siello S leads.
Arm/Group | BIOTRONIK Siello S Lead
Number analyzed (Participants) | 538
percentage of participants | 100 [99.3 to 100]
Statistical Analysis 1: Comparison: BIOTRONIK Siello S Lead; The primary endpoint 3 hypothesis was evaluated by performing an exact, binomial test comparing a binomial proportion (successful sensing and pacing rate at 12 months) to 97.0%, with Type I error (alpha) or 0.025 and power of 80%; Test type: Superiority; p < 0.0001, Exact, binomial

4. Primary Outcome: Ventricular Siello S Lead Safety at 5 Years
Description: The overall percentage of subjects with adverse events that require additional invasive intervention to resolve, related to the Siello leads implanted in the ventricle with a BIOTRONIK Evia pacemaker device through 5 years follow-up. This was evaluated as an adverse event free-rate (AEFR).
Time Frame: 5-Years
Population: The Post-Market cohort included all patient who were enrolled in the study and had a Siello lead implanted in the right ventricular position.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- BIOTRONIK Siello S Ventricular Lead: Patients with a BIOTRONIK pacemaker system including a Siello S ventricular lead.
Arm/Group | BIOTRONIK Siello S Ventricular Lead
Number analyzed (Participants) | 1728
percentage of participants | 99.71 [99.33 to 99.91]
Statistical Analysis 1: Comparison: BIOTRONIK Siello S Ventricular Lead; The primary endpoint 4 hypothesis was evaluated by performing an exact, binomial test comparing a binomial proportion (AEFR at 5 years) to 92.5%, with Type I error (alpha) or 0.025 and power of 80%; Test type: Superiority; On April 15, 2019, BIOTRONIK received FDA approval to transition the ongoing SIELLO Post Approval Registry to a new EP PASSION real-world data methodology. As of study closure, the number of subjects with complete data required to perform the hypothesis test was not met. Therefore, this outcome measure was not analyzed

5. Primary Outcome: Ventricular Siello S Lead Safety at 5 Years - Individual Adverse Event Rates
Description: Evaluation of the individual adverse events contributing to the outcome measure 'Ventricular Siello S Lead Safety at 5 Years'.
Time Frame: 5-years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIOTRONIK Siello S Ventricular Lead
Number analyzed (Participants) | 1728
percentage of participants
  Lead impedance out of range, High | 0.17 [0.04 to 0.51]
  Lead conductor fracture | 0.12 [0.01 to 0.42]

6. Secondary Outcome: Atrial Siello S Lead Safety at 5 Years
Description: The overall percentage of subjects with adverse events that require additional invasive intervention to resolve, related to the Siello leads implanted in the atrium with a BIOTRONIK Evia pacemaker device through 5 years follow-up. This was evaluated as an adverse event free-rate (AEFR).
Time Frame: 5-years
Population: The Post-Market cohort included all patient who were enrolled in the study and had a Siello lead implanted in the right atrial position.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- BIOTRONIK Siello S Atrial Lead: Patients with a BIOTRONIK pacemaker system including Siello S atrial lead.
Arm/Group | BIOTRONIK Siello S Atrial Lead
Number analyzed (Participants) | 1493
percentage of participants | 99.87 [99.52 to 99.98]

7. Secondary Outcome: Atrial Siello S Lead Safety at 5 Years - Individual Adverse Event Rates
Description: Evaluation of the individual adverse events contributing to the outcome measure 'Atrial Siello S Lead Safety at 5 Years'.
Time Frame: 5-years
Population: On April 15, 2019, BIOTRONIK received FDA approval to transition the ongoing SIELLO Post Approval Registry to a new EP PASSION real-world data methodology. Therefore, this outcome measure was not completed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIOTRONIK Siello S Atrial Lead
Number analyzed (Participants) | 1493
percentage of participants
  Intermittent capture | 0.07 [0.01 to 0.37]
  Suspected lead failure | 0.07 [0.01 to 0.37]

8. Secondary Outcome: Pacing Threshold Measurements for Siello S Leads at 12 Months
Description: Pacing threshold measurements for Siello S leads implanted in the atrium or ventricle at the 12 month follow-up visit.
Time Frame: 12-months
Population: All originally implanted ventricular or atrial Siello leads with 12-month follow-up data entered into the EDC on or before April 3, 2015 are included in this analysis.
Measure: Mean (Standard Deviation); unit: volts
Groups:
- Siello S Ventricular Leads: All originally implanted ventricular Siello leads with 12-month follow-up data entered into the EDC on or before April 3, 2015 are included in this analysis. For data poolability, thresholds performed with a pulse-width of 0.4 or 0.5 ms were requested. Only data collected at 0.4 or 0.5 ms pulse-width was analyzed and reported.
- Siello S Atrial Leads: All originally implanted atrial Siello leads with 12-month follow-up data entered into the EDC on or before April 3, 2015 are included in this analysis. For data poolability, thresholds performed with a pulse-width of 0.4 or 0.5 ms were requested. Only data collected at 0.4 or 0.5 ms pulse-width was analyzed and reported.
Arm/Group | Siello S Ventricular Leads | Siello S Atrial Leads
Number analyzed (Participants) | 505 | 389
volts | 0.86 (0.29) | 0.85 (0.35)

9. Secondary Outcome: Sensing Measurements for Siello S Leads at 12 Months
Description: Sensing measurements for Siello S leads implanted in the atrium or ventricle at the 12 month follow-up visit.
Time Frame: 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Siello S Ventricular Leads: All originally implanted ventricular Siello leads with 12-month follow-up data entered into the EDC on or before April 3, 2015 are included in this analysis.
- Siello S Atrial Leads: All originally implanted atrial Siello leads with 12-month follow-up data entered into the EDC on or before April 3, 2015 are included in this analysis.
Arm/Group | Siello S Ventricular Leads | Siello S Atrial Leads
Number analyzed (Participants) | 446 | 429
mV | 12.68 (5.02) | 3.66 (1.92)

10. Secondary Outcome: Impedance Measurements for Siello S Leads at 12 Months
Description: Impedance measurements for Siello S leads implanted in the atrium or ventricle at the 12 month follow-up visit.
Time Frame: 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | Siello S Ventricular Leads | Siello S Atrial Leads
Number analyzed (Participants) | 515 | 441
Ohms | 595.7 (89.1) | 524.0 (66.7)

11. Secondary Outcome: Percentage of Participants With Other Adverse Events
Description: The overall percentage of subjects with reportable adverse events that were excluded from primary and secondary objectives and occurred through 5 years of follow-up. This was evaluated as an adverse event free-rate (AEFR). Adverse events were considered reportable if the event was related to the implant procedure, implanted pulse generator, or implanted leads.
Time Frame: 5-years
Population: The Post-Market cohort included all patient who were enrolled in the study and had one or two Siello leads implanted.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIOTRONIK Siello S Lead
Number analyzed (Participants) | 1758
percentage of participants | 84.02 [82.22 to 85.70]

12. Secondary Outcome: Siello S Lead Effectiveness at 5 Years
Description: Success rate of the implanted system to deliver long-term pacing at 5-years post-implant.
Time Frame: 5-years
Population: The Post-Market cohort included all patient who were enrolled in the study and had one or two Siello leads implanted.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIOTRONIK Siello S Lead
Number analyzed (Participants) | 1758
percentage of participants | 99.94 [99.68 to 99.99]

13. Secondary Outcome: Pacing Threshold Measurements for Siello S Leads Through 5 Years
Description: Pacing threshold measurements for Siello S leads implanted in the atrium or ventricle through 5 years of follow-up.
Time Frame: 5-years
Population: All originally implanted ventricular or atrial Siello leads with implant and follow-up data entered into the EDC on or before April 17, 2019 are included in this analysis.
Measure: Mean (Standard Deviation); unit: volts
Groups:
- Siello S Ventricular Leads: All originally implanted ventricular Siello leads with follow-up data entered into the EDC on or before April 17, 2019 are included in this analysis. For data poolability, thresholds performed with a pulse-width of 0.4 or 0.5 ms were requested. Only data collected at 0.4 or 0.5 ms pulse-width was analyzed and reported.
- Siello S Atrial Leads: All originally implanted atrial Siello leads with follow-up data entered into the EDC on or before April 17, 2019 are included in this analysis. For data poolability, thresholds performed with a pulse-width of 0.4 or 0.5 ms were requested. Only data collected at 0.4 or 0.5 ms pulse-width was analyzed and reported.
Arm/Group | Siello S Ventricular Leads | Siello S Atrial Leads
Number analyzed (Participants) | 1727 | 1493
volts | 0.84 (0.34) | 0.83 (0.34)

14. Secondary Outcome: Sensing Measurements for Siello S Leads Through 5 Years
Description: Sensing measurements for Siello S leads implanted in the atrium or ventricle through the 5 year follow-up visit.
Time Frame: 5-years
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Siello S Ventricular Leads: All originally implanted ventricular Siello leads with follow-up data entered into the EDC on or before April 17, 2019 are included in this analysis.
- Siello S Atrial Leads: All originally implanted atrial Siello leads with follow-up data entered into the EDC on or before April 17, 2019 are included in this analysis.
Arm/Group | Siello S Ventricular Leads | Siello S Atrial Leads
Number analyzed (Participants) | 1727 | 1493
mV | 12.17 (4.60) | 3.53 (1.95)

15. Secondary Outcome: Impedance Measurements for Siello S Leads Through 5 Years
Description: Impedance measurements for Siello S leads implanted in the atrium or ventricle through the 5 year follow-up visit.
Time Frame: 5-years
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | Siello S Ventricular Leads | Siello S Atrial Leads
Number analyzed (Participants) | 1727 | 1493
Ohms | 597.6 (100.0) | 514.4 (72.6)

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: According to the study protocol, sites were required to report all patient deaths and all adverse events that were considered related to the implant procedure, implanted pulse generator, or implanted leads. Adverse events determined to be not related to the implant procedure, implanted pulse generator, or implanted leads were not collected.
  Reported adverse events were defined as a serious or 'other' adverse event according to the clinicaltrials.gov definition.
Arm/Group | BIOTRONIK Siello S Lead
All-Cause Mortality (participants affected / at risk) | 356/1758
Serious Adverse Events (participants affected / at risk) | 145/1758
Other Adverse Events (participants affected / at risk) | 154/1758
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOTRONIK Siello S Lead (N=1758)
Accumulation of serous fluid in pocket (Cardiac disorders) | 1 (1)
Cardiac perforation associated with the RA lead (Cardiac disorders) | 4 (4)
Cardiac perforation associated with the RV lead (Cardiac disorders) | 3 (4)
Cardiac perforation associated with the Siello lead (Cardiac disorders) | 1 (1)
Inability to place RA lead (Cardiac disorders) | 1 (1)
Lead related thrombosis (Cardiac disorders) | 1 (1)
LV lead related extracardiac stimulation (Cardiac disorders) | 2 (2)
LV lead related lead dislodgement (Cardiac disorders) | 2 (2)
Pulse generator failure (Cardiac disorders) | 1 (1)
Pulse generator migration (Cardiac disorders) | 1 (1)
RA lead related (non-Siello) lead dislodgement (Cardiac disorders) | 1 (1)
RA lead related high pacing threshold (Cardiac disorders) | 2 (2)
RA lead related lead dislodgement (Cardiac disorders) | 39 (41)
RA lead suspected lead failure (Cardiac disorders) | 1 (1)
RA lead undersensing or loss of sensing (Cardiac disorders) | 1 (1)
RV lead conductor fracture (Cardiac disorders) | 2 (2)
RV lead impedance out of range, high impedance (Cardiac disorders) | 3 (3)
RV lead intermittent capture, no lead capture (Cardiac disorders) | 3 (3)
RV lead lead insulation failure (Cardiac disorders) | 1 (1)
RV lead related (non-Siello) lead dislodgement (Cardiac disorders) | 1 (1)
RV lead related extracardiac stimulation (Cardiac disorders) | 1 (1)
RV lead related high pacing threshold (Cardiac disorders) | 5 (5)
RV lead related lead dislodgement (Cardiac disorders) | 22 (23)
Software malfunction (Cardiac disorders) | 1 (1)
Twiddler's syndrome (General disorders) | 5 (5)
Implant procedure related infection (Infections and infestations) | 14 (16)
Prosthetic aortic valve endocarditis (Infections and infestations) | 1 (1)
Secondary infection (Infections and infestations) | 2 (2)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac perforation (Surgical and medical procedures) | 2 (2)
Damage to lead during procedure (Surgical and medical procedures) | 6 (6)
Hematoma (Surgical and medical procedures) | 9 (10)
Lead dislodgement during a procedure (Surgical and medical procedures) | 4 (5)
Lead reversed in header (Surgical and medical procedures) | 1 (1)
Loose set-screw (Surgical and medical procedures) | 6 (6)
Pneumothorax (Surgical and medical procedures) | 8 (8)
Pocket pain (Surgical and medical procedures) | 6 (8)
Possible transient ischemic attack (Surgical and medical procedures) | 1 (1)
Pulmonary embolism (Surgical and medical procedures) | 2 (2)
Respiratory arrest (Surgical and medical procedures) | 1 (1)
Respiratory distress (Surgical and medical procedures) | 1 (1)
Venous occlusion (Surgical and medical procedures) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOTRONIK Siello S Lead (N=1758)
Atrial oversensing (Cardiac disorders) | 1 (1)
Cardiac perforation associated with the LV lead (Cardiac disorders) | 1 (1)
Cardiac perforation associated with the RV lead (Cardiac disorders) | 1 (1)
Cardiac perforation associated with the Siello lead (Cardiac disorders) | 1 (1)
Failure of fixation helix to retract (Cardiac disorders) | 1 (1)
Inability to place LV lead (Cardiac disorders) | 1 (1)
LV lead impedance out of range, high impedance (Cardiac disorders) | 1 (1)
LV lead intermittent capture, no lead capture (Cardiac disorders) | 1 (1)
LV lead related diaphragmatic stimulation (Cardiac disorders) | 1 (1)
LV lead related extracardiac stimulation (Cardiac disorders) | 15 (16)
LV lead related high pacing threshold (Cardiac disorders) | 11 (12)
LV lead related lead dislodgement (Cardiac disorders) | 3 (3)
LV lead related oversensing (Cardiac disorders) | 1 (1)
RA lead (non-Siello) undersensing or loss of sensing (Cardiac disorders) | 2 (2)
RA lead intermittent capture, no lead capture (Cardiac disorders) | 1 (1)
RA lead related (non-Siello) high pacing threshold (Cardiac disorders) | 1 (1)
RA lead related extracardiac stimulation (Cardiac disorders) | 1 (1)
RA lead related high pacing threshold (Cardiac disorders) | 12 (12)
RA lead related lead dislodgement (Cardiac disorders) | 3 (3)
RA lead undersensing or loss of sensing (Cardiac disorders) | 11 (11)
RV lead impedance out of range, high impedance (Cardiac disorders) | 3 (3)
RV lead related (non-Siello) high pacing threshold (Cardiac disorders) | 1 (1)
RV lead related extracardiac stimulation (Cardiac disorders) | 2 (2)
RV lead related high pacing threshold (Cardiac disorders) | 14 (14)
RV lead related lead dislodgement (Cardiac disorders) | 1 (1)
RV lead undersensing or loss of sensing (Cardiac disorders) | 5 (6)
Transient inhibition secondary to EMI (Cardiac disorders) | 1 (1)
Implant procedure related infection (Infections and infestations) | 19 (19)
Allergic reaction at pocket site (Surgical and medical procedures) | 1 (1)
Damage to lead during procedure (Surgical and medical procedures) | 1 (1)
Hematoma (Surgical and medical procedures) | 30 (30)
Inability to place LV lead (Surgical and medical procedures) | 1 (1)
Inability to place RA lead (Surgical and medical procedures) | 2 (2)
Inability to place RV lead (Surgical and medical procedures) | 1 (1)
Pericardial effusion (Surgical and medical procedures) | 1 (1)
Pericarditis (Surgical and medical procedures) | 1 (1)
Pleural effusion (Surgical and medical procedures) | 1 (1)
Pneumothorax (Surgical and medical procedures) | 2 (2)
Pocket pain (Surgical and medical procedures) | 7 (7)
RA lead dislodgement during a procedure (Surgical and medical procedures) | 1 (1)
Venous occlusion (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT01791127/Prot_SAP_000.pdf